CLINICAL TRIAL: NCT06946576
Title: Infant Survival and Long-term Outcomes Following Fetoscopic Endoluminal Tracheal Occlusion in Severe Left and Right Congenital Diaphragmatic Hernia, A Phase III Trial
Brief Title: Safety and Efficacy of Fetoscopic Endoluminal Tracheal Occlusion in Congenital Diaphragmatic Hernia
Status: Not yet recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Oregon Health and Science University (Other)
Responsible Party: Principal Investigator, Raphael Sun, Principal Investigator, Oregon Health and Science University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: STUDY00027320
Record Dates: First submitted 2025-03-18; First posted 2025-04-27 (Actual); Last update posted 2025-09-02 (Actual); Status verified 2025-08

CONDITIONS: Congenital Diaphragmatic Hernia
Keywords: Fetal Surgery; Fetoscopic Endoluminal Tracheal Occlusion (FETO)
MeSH Terms: conditions — Hernias, Diaphragmatic, Congenital

STUDY DESIGN:
Intervention Model Description: Unblinded non-randomized double-arm phase III study
Masking Description: This is an unblinded trial
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Fetal treatment arm (Experimental): Cases that will undergo Fetoscopic Endoluminal Tracheal Occlusion (FETO) procedure.
  Interventions: Device: Fetoscopic Endoluminal Tracheal Occlusion (FETO) Procedure
- Expectant management arm (No Intervention): Cases that meet study inclusion criteria but voluntarily decline the Fetoscopic Endoluminal Tracheal Occlusion (FETO) procedure. These cases will undergo the standard of clinical care.

INTERVENTIONS:
Device: Fetoscopic Endoluminal Tracheal Occlusion (FETO) Procedure — FETO procedure involves insertion of a balloon into the fetal trachea under IV sedation with local anesthesia or combined spinal-epidural anesthesia. Balloon removal will take place up to 7 weeks after insertion.
  Other Names: FETO; GoldBAL2 Detachable Balloon
  Arms: Fetal treatment arm

SUMMARY:
The purpose of this study is to evaluate the safety and efficacy of Fetoscopic Endoluminal Tracheal Occlusion (FETO) in cases of severe Congenital Diaphragmatic Hernia (CDH).

DETAILED DESCRIPTION:
This is an un-blinded, non-randomized, double-arm phase III clinical trial designed to evaluate the safety and efficacy of Fetoscopic Endoluminal Tracheal Occlusion in cases of severe Congenital Diaphragmatic Hernia (CDH) and intrathoracic liver herniation. Patients in the intervention arm will undergo balloon insertion into the fetal trachea between 27 and 30 weeks of gestation. Fetoscopic removal of the balloon occlusion will be performed at 34 weeks gestation.

ELIGIBILITY:
Inclusion Criteria:

* Pregnant person age 18 years or older
* Singleton pregnancy
* Normal fetal karyotype with confirmation by culture results, Chromosomal Microarray (CMA) with non-pathological variants, Whole Exome Sequencing (WES) or Whole Genome Sequencing (WGS). Results by florescence in situ hybridization (FISH) will be acceptable if the patient is >26 weeks gestation
* Gestational age at enrollment less than 29 weeks 6 days
* Intrathoracic liver herniation
* Isolated left Congenital Diaphragmatic Hernia (CDH) with Lung to Head Circumference Ratio (LHR) <30% at enrollment OR isolated right CDH with LHR <= 45% at enrollment
* Cervical length by transvaginal ultrasound >= 20 mm within 24 hours of FETO procedure
* Psychosocial criteria
* Able to provide informed consent

Exclusion Criteria:

* Patient < 18 years of age
* Multi-fetal pregnancy
* History of natural rubber latex allergy
* Preterm labor, cervix shortened (<20 mm at enrollment or within 24 hours of FETO balloon insertion procedure) or uterine anomaly strongly predisposing to preterm labor or placenta previa
* Psychosocial ineligibility precluding consent
* Inability to reside within 30 minutes of OHSU
* Inability to comply with the travel for the follow-up requirements of the trial
* Lack of a support person (e.g., spouse, partner, mother) available to stay with the patient for the duration of the pregnancy at OHSU.
* Bilateral CDH, isolated left sided CDL with LHR >= 30% or isolated right side CDH with LHR >45% as determined by ultrasound
* No intrathoracic liver herniation
* Additional fetal anomaly and chromosomal abnormalities, associated anomalies recognized to alter survival prognosis (i.e. congenital heart disease) or presence of an underlying genetic syndrome (i.e. Fryns) by ultrasound, MRI, or echocardiogram at the fetal treatment center
* Maternal contraindication to fetoscopic surgery or severe maternal medical condition in pregnancy
* History of incompetent cervix with or without cerclage
* Placental abnormalities (previa, abruption, accreta) known at time of enrollment
* Maternal-fetal Rh isoimmunization, Kell sensitization or neonatal alloimmune thrombocytopenia affecting the current pregnancy
* Maternal HIV, Hepatitis-B, Hepatitis-C status positive because of the increased risk of transmission to the fetus during maternal-fetal surgery. If the patient's HIV or Hepatitis status is unknown, the patient must be tested and found to have negative results before enrollment
* Uterine anomaly such as large or multiple fibroids or Mullerian duct abnormality
* No safe or technically feasible fetoscopic approach to balloon placement
* Participation in another intervention study that influences maternal and fetal morbidity and mortality or participation in this trial in a previous pregnancy.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2025-09 (Estimated); Primary Completion 2030-04 (Estimated); Study Completion 2030-04 (Estimated)

PRIMARY OUTCOMES:
Outcomes of placement and removal of FETO device | Device placement will take place between 27 weeks 0 days and 29 weeks 6 days gestation. Removal will take place between 34 weeks 0 days and 34 weeks 6 days.
  Whether placement and removal of the FETO device was successful or not
Compare survival to discharge between FETO and expectant management | Evaluated upon discharge from the NICU (typically 6 months to 1 year after birth)
  Evaluate rates of survival to discharge from the neonatal intensive care units (NICU) between fetuses treated with the FETO and those undergoing expectant management
FETO Complications | Information about adverse events and complications will take place from study enrollment (gestational age less than 29 weeks) to study conclusion (24 months post-birth)
  Evaluate the frequency of maternal and fetal complications associated with the FETO procedure

SECONDARY OUTCOMES:
Long-term mortality and morbidities | 6 months, 12 months, 18 months, and 24 months of age
  Comparison of rates of long-term mortality and morbidities compared between FETO group and those who underwent expectant management.

CONTACTS AND LOCATIONS:
Overall Officials: Raphael Sun, MD, Principal Investigator — Oregon Health and Science University; Andrew Chon, MD, Principal Investigator — Oregon Health and Science University
Locations (1):
- Oregon Health & Science University, Portland, Oregon, United States